CLINICAL TRIAL: NCT05436691
Title: The Effect of Information and Coping With Anxiety Training Given to Women Before Hysterectomy on Their Level of Anxiety: A Post-Test Randomized Controlled Experimental Study
Brief Title: The Effect of Information and Coping With Anxiety Training Given to Women Before Hysterectomy on Their Level of Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elcin Alacam, MSc, Nurse, Principal Investigator, Mersin Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinCity
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Hysterectomy; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information and Coping with Anxiety Training Intervention (Experimental): The intervention group received information and coping with anxiety training by an instructor.
  Interventions: Other: Information and Coping with Anxiety Training
- Control (No Intervention): No intervention was applied to the control group.Data were collected from the control group simultaneously with the study group.

INTERVENTIONS:
Other: Information and Coping with Anxiety Training — Informing and Coping with Anxiety Training was given to the experimental group before the operation through a prepared booklet.The information booklet about the training was created by the researchers by reviewing the current literature. The booklet provides information for patients scheduled for hysterectomy about how to cope with surgery-related anxiety. The booklet provides information on what the hysterectomy is, why it is performed, what risks it has, what should be done before, during and after the hysterectomy, what rules the patient should comply with after hysterectomy, in which cases she should present to the health institution, what changes she might experience in her social, physical, sexual and emotional life after the surgery. The booklet also provides information about discharge training and coping with anxiety.
  Arms: Information and Coping with Anxiety Training Intervention

SUMMARY:
Purpose: In this study, it was aimed to determine the effect of information and coping with anxiety training given to women before they undergo hysterectomy on their anxiety levels.

Design and Methods: The parallel group post-test randomized controlled experimental design was used in the study. The study sample comprised 59 women.

ELIGIBILITY:
Inclusion Criteria:

* agreeing to participate in the study,
* being able to speak and understand Turkish,
* being in the age group of 18-65 years,
* being admitted to the aforementioned clinic with a planned hysterectomy surgery,
* not having any health problems preventing the person from hearing and speaking,
* being conscious, being oriented and cooperated,
* not having received any training on hysterectomy before the surgery and during discharge.

Exclusion Criteria:

* not agreeing to participate in the study,
* not being able to speak and understand Turkish,
* being under the age group of 18 years,
* not being admitted to the aforementioned clinic with a planned hysterectomy surgery,
* having any health problems preventing the person from hearing and speaking,
* not being conscious, being oriented and cooperated,
* having received any training on hysterectomy before the surgery and during discharge.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — being a woman depending on the hysterectomy surgery
Enrollment: 59 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Anxiety was assessed using the State-Trait Anxiety Scale. | preoperative
  The total score obtained from both scales varies between 20 and 80. It states that 0-19 points mean no anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-79 points mean severe anxiety, and individuals with a score of 60 and above need professional help

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No